CLINICAL TRIAL: NCT00841347
Title: Sleep and Obesity in Teenagers: Impact of Sleep Length and Quality on Obesity and Diabetes Risks in Teenagers.
Brief Title: Sleep and Obesity in Teenagers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 2008.525
Record Dates: First submitted 2009-02-10; First posted 2009-02-11 (Estimated); Last update posted 2017-08-03 (Actual); Status verified 2017-08

CONDITIONS: Obesity
Keywords: Obesity; Glucose metabolism disorders; Appetite regulation; Sleep; Adolescent; Randomized controlled trials
MeSH Terms: conditions — Obesity; Glucose Metabolism Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (No Intervention): Study of habitual sleep length on non obese teen group
- 2 (Experimental): Study of habitual sleep length period followed by extended sleep length period on obese teen group
  Interventions: Behavioral: habitual sleep length period + extended sleep length period
- 3 (Experimental): Study of extended sleep length period followed by habitual sleep length period on obese teen group
  Interventions: Behavioral: extended sleep length period + habitual sleep length period

INTERVENTIONS:
Behavioral: habitual sleep length period + extended sleep length period — On obese group, realisation of an habitual sleep length period followed by an extended sleep length period
  Arms: 2
Behavioral: extended sleep length period + habitual sleep length period — On obese group, realisation of an extended sleep length period followed by an habitual sleep length period
  Arms: 3

SUMMARY:
This study aims to investigate

1. whether sleep extension results in improvements of endocrine and metabolic markers of obesity and diabetes in obese teenagers,
2. the relationship between habitual sleep quality and duration and markers of obesity and diabetes in lean and obese teenagers.

DETAILED DESCRIPTION:
Inclusion of 13 obese teens. Duration : 1 week of screening period + 1 week of intervention: habitual/extended sleep length + 1 week of intervention: extended/habitual sleep length. A wash out period of at least 3 months will be required between the two interventions.

Inclusion of 13 non obese healthy teen controls for measuring reference sleep duration and physiology level. Duration for these group: 1 week of screening period + 1 week of habitual sleep length

ELIGIBILITY:
Inclusion Criteria:

* Male or female over 15 and under 18 year-old.
* Teenager with normal weight or stage 2 obesity, according to international standards (WHO)
* Post-pubescent teenagers (menstruation for girls and stage 4-5 of Tanner scale for boys)
* Teens with an social security
* Girl with negative urine pregnancy test

Exclusion Criteria:

* Active smoker (interview)
* Refuse consent (parents or teen)
* Addiction such as coffee, drug…(interview)
* Medicinal treatment that may influence sleep and measured variables (interview)
* Obesity diagnosis : less than 1 year (interview)
* Concomitant diseases : renal or hepatic failure, iron deficit, diabetes, endocrinal pathology, hypertension
* Anxiety (Spielberg>56), , depression (CDI>19).
* Mild or sever insomnia (ISI>15), poor sleep quality (PSQI >10), excessive sleepiness (Epworth>10, sleep) length>9 hour), extreme circadian typology (Horne et Ostberg from 70 to 86 or 16 to 30)
* Blood sample taken within the last two months before inclusion
* Mild or severe sleep apnoea or excessive leg movements according to EEG analysis

Ages: 15 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 41 (Actual)
Dates: Start 2009-02; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
The influence of sleep extension on leptin level for the obese teens group. | at the end of each sleep experimental period

SECONDARY OUTCOMES:
Difference between the two groups (obese vs non-obese) regarding sleep length and delta waves activity. | during each sleep experimental period (habitual or extended)
Study the correlation between delta waves activity and habitual sleep length | During each sleep experimental period
Study the correlation between delta waves activity and psychological, behavioural, anthropometric and physiological markers of obesity and its co morbidities | During each sleep experimental period

CONTACTS AND LOCATIONS:
Overall Officials: Karine SPIEGEL, PhD, Study Chair — Institut National de la Santé Et de la Recherche Médicale, France; Behrouz KASSAI, MD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hospices Civils de Lyon, Lyon, France